CLINICAL TRIAL: NCT03688347
Title: The Role of Microbiome in Lung Cancer and Other Malignancies
Brief Title: Microbiome in Lung Cancer and Other Malignancies
Status: Completed | Type: Observational
Sponsor: Taher Abu Hejleh (Other)
Collaborators: Holden Comprehensive Cancer Center (Other); Iowa Institute of Human Genetics (Unknown)
Responsible Party: Sponsor-Investigator, Taher Abu Hejleh, Clinical Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 201712819
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Lung Cancer; Cancer; Malignancy
MeSH Terms: conditions — Lung Neoplasms; Neoplasms | interventions — Gene Library

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bacterial DNA will be isolated from oral, skin, and nasal swabs, as well as stool samples. The extracted DNA will be subsequently used for microbiome analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Nasal Swab — The swab is removed from packaging, moistened with sterile water if needed to prevent any discomfort to the participant. The swab is gently inserted less than one inch into the anterior nare (nostril) until resistance is met at turbinate. Then it is rotated several times against nasal wall and repeated in other nostril using the same swab.
Procedure: Oral Swab — The swab is removed from packaging, moistened with sterile water if needed to prevent any discomfort to the participant. The swab is gently rubbed along the inside of the participant's cheek for 5-10 seconds.
Other: Stool Collection — A stool collection kit will be sent home with each participant. It will include instructions on how to collect the stool specimen and how to return the kit.
Genetic: Microbiome analysis — Study of microbial communities found in and on the human body.
Genetic: DNA Banking — Secure, long term storage of an individual's genetic material.
Procedure: Skin Swab — Gentle rubbing of the swab will be applied to the skin on the dorsal part of the hand.

SUMMARY:
To characterize the fecal, skin, nasal and oral microbiome and metabolome in patients with lung cancer and other malignancies, and correlate to treatment response and toxicities of various therapies including immunotherapy, chemotherapy and targeted therapy, etc.

DETAILED DESCRIPTION:
Patients will be asked to provide nasal, oral and skin swabs, as well as stool samples during their regular clinic visits, at the baseline before desired therapy is given, and at the time when treatment is changed due to either disease progression or unbearable toxicities leading to treatment stop/change. If treatment stop/held is due to toxicities, a 3rd set of samples will be collected when toxicities reduce to less than grade 1. The samples will be subjected to DNA extraction followed by 16S rRNA and/or shotgun sequencing metagenomic analysis. The data will be correlated to clinical response from treatments, toxicities, clinical data (use of antibiotics, PPIs, lab parameters, etc.) and tissue genetic/immunological characteristics (mutations, PDL1 expression, etc.) for review of response. This is not data to be used for treatment of these subjects.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with lung cancer and other malignancies who are candidates for systemic therapies such as immunotherapy and chemotherapy

Eligibility criteria for studying microbiome in patients receiving immunotherapy:

* Patients with advanced/recurrent lung cancer (including both NSCLC and SCLC) and other solid tumors of our study interest (e.g. GU cancer and melanoma, etc.) that initiate a new line of immunotherapy (can be 1st or later line), either alone or in combination with chemotherapy, targeted therapy or other immunotherapy.
* Patients can be in other clinical trials as long as they meet criteria 1.
* Prior treatment with immunotherapy is acceptable as long as criteria 1 is met. For example, a new line therapy with pembrolizumab plus pemetrexed after failing pembrolizumab is considered eligible.
* Patients who are to start immunotherapy maintenance after chemoradiation therapy are eligible (e.g. NSCLC patients who will be on durvalumab maintenance)
* Patients who are to start immunotherapy after local therapies (e.g. radiation, ablation, etc.) are eligible.
* Immunotherapy must have component of anti-PD-1/PD-L1 agents (e.g. nivolumab, pembrolizumab, atezolizumab, durvalumab and avelumab, etc.) or anti-CTLA4 (e.g. ipilimumab)

Exclusion Criteria:

* Patients < 18 years of age
* Patients that are pregnant
* Patients taking more than 2 alcoholic drinks per day and those using non-medical drugs such as marijuana, cocaine, heroine, etc.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All individuals, meeting eligibility requirements will be eligible to participate in the study by providing samples during times of routine care for lung cancer and other malignancies.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2022-05-09 (Actual)

PRIMARY OUTCOMES:
Identify and compare bacteria within given samples through standard protocol and 16S rRNA amplicon | Time of study enrollment up to one year
  Bacterial DNA will be isolated from stool/swab samples using standard protocol. Fecal micobiota will be examined based on an 16S rRNA amplicon.

SECONDARY OUTCOMES:
Correlate data from samples with patient clinical information | Time of study enrollment up to one year
  Correlate data from samples with patient clinical information regarding overall response rates.
Number of treatment related adverse events (AE) as defined by National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 | Time of study enrollment up to one year
  Record from each clinical visit the AEs from immunotherapy or its combination with chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Taher Abu Hejleh, MBBS, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Strouse C, Mangalam A, Zhang J. Bugs in the system: bringing the human microbiome to bear in cancer immunotherapy. Gut Microbes. 2019;10(2):109-112. doi: 10.1080/19490976.2018.1511665. Epub 2018 Sep 5. PMID 30183502
- [Background] Swami U, Zakharia Y, Zhang J. Understanding Microbiome Effect on Immune Checkpoint Inhibition in Lung Cancer: Placing the Puzzle Pieces Together. J Immunother. 2018 Oct;41(8):359-360. doi: 10.1097/CJI.0000000000000232. PMID 29781826
- [Derived] Chau J, Yadav M, Liu B, Furqan M, Dai Q, Shahi S, Gupta A, Mercer KN, Eastman E, Hejleh TA, Chan C, Weiner GJ, Cherwin C, Lee STM, Zhong C, Mangalam A, Zhang J. Prospective correlation between the patient microbiome with response to and development of immune-mediated adverse effects to immunotherapy in lung cancer. BMC Cancer. 2021 Jul 13;21(1):808. doi: 10.1186/s12885-021-08530-z. PMID 34256732